CLINICAL TRIAL: NCT06111053
Title: Harm Reduction in Smokers With Obesity: Impact of Contingent Incentives and E-Cigarettes
Brief Title: Trial for Harm Reduction With Incentives & Vaping E-cigarettes
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2022003359; P20GM130414 (NIH)
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Smoking Cessation
Keywords: obesity; overweight; electronic nicotine delivery systems; contingent incentives; harm reduction
MeSH Terms: conditions — Obesity; Smoking Cessation; Overweight; Vaping; Harm Reduction | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: A 2x2 factorial design comparing
  * contingent incentives (CI) for smoking abstinence to noncontingent incentives (NI)
  * the provision of ENDS (ENDS) to no provision of ENDS (No ENDS)
  SWO (N=36) will be randomized to receive 4 weeks of monetary incentives contingent on their smoking abstinence (CI) or after completing breath samples only (NI). They will also be randomized to receive either a 6-week provision of ENDS with information communicating the comparative risk of ENDS use relative to smoking or information communicating the comparative risk of ENDS relative to smoking without ENDS provision. Conditions are as follows:
  * C1: ENDS + CI
  * C2: NoENDS + CI
  * C3: ENDS + NI
  * C4: NoENDS + NI
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will not know the outcome of randomized assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ENDS and CI (Experimental): Participants in this arm will receive information about the comparative risk of electronic nicotine delivery systems (ENDS) relative to smoking as well as 6 weeks' worth of provisions of ENDS and will receive 4 weeks of monetary incentives for complete abstinence from smoking (after a controlled ramp down of smoking).
  Interventions: Other: ENDS; Other: CI
- No ENDS and CI (Experimental): Participants in this arm will receive information about the comparative risk of electronic nicotine delivery systems (ENDS) relative to smoking and will receive 4 weeks of monetary incentives for complete abstinence from smoking (after a controlled ramp down of smoking).
  Interventions: Other: CI; Other: No ENDS
- ENDS and NI (Experimental): Participants in this arm will receive information about the comparative risk of electronic nicotine delivery systems (ENDS) relative to smoking as well as 6 weeks' worth of provisions of ENDS and will receive monetary incentives for providing breath samples only (non-contingent on smoking status).
  Interventions: Other: ENDS; Other: NI
- No ENDS and NI (Experimental): Participants in this arm will receive information about the comparative risk of electronic nicotine devices (ENDs) relative to smoking and will receive monetary incentives for providing breath samples only (non-contingent on smoking status).
  Interventions: Other: No ENDS; Other: NI

INTERVENTIONS:
Other: ENDS — Participants in active comparator groups that include ENDS will receive 6-weeks worth of ENDS supplies.
  Other Names: Electronic Nicotine Delivery Systems
  Arms: ENDS and CI; ENDS and NI
Other: CI — Participants in active comparator groups will receive incentives that vary based on participant abstinence from smoking, measured by a carbon monoxide breath sample.
  Other Names: Contingent Incentives
  Arms: ENDS and CI; No ENDS and CI
Other: No ENDS — Participants in active comparator groups labeled No ENDS will only receive information about the comparative risk of ENDS relative to combustible cigarettes.
  Arms: No ENDS and CI; No ENDS and NI
Other: NI — Participants in active comparator groups labeled NI will receive compensation for each breath sample provided throughout the study, with no variation.
  Other Names: Non-Contingent Incentives
  Arms: ENDS and NI; No ENDS and NI

SUMMARY:
The purpose of this study is to provide preliminary information on the effect of electronic nicotine delivery systems (ENDS) provisions and contingent incentives (CI) on smoking in individuals with overweight/obesity who smoke cigarettes (SWO). All participants will be provided information on the comparative risk of ENDS relative to cigarette smoking, and a randomized group of participants will be provided ENDS provisions for 6 weeks. All participants will complete breath samples for 28 days to measure their exhaled carbon monoxide and will either receive fixed incentives for sample completion or receive varying incentives contingent on their carbon monoxide levels. Researchers will compare groups to understand the effect of each condition on smoking-related behavior.

DETAILED DESCRIPTION:
Individuals with overweight/obesity who smoke cigarettes (SWO) have greatly increased risks of metabolic, cardiac, and pulmonary diseases due to the synergistic effects of tobacco and obesity. Switching to electronic nicotine delivery systems (ENDS) may decrease the risk of negative health outcomes and be a promising approach for SWO. The purpose of this study is to provide preliminary information on the effect of electronic nicotine delivery systems (ENDS) provisions and contingent incentives (CI) on individuals with overweight/obesity who smoke cigarettes (SWO). The primary aim of this study is to examine the effect of ENDS provision on smoking and the effect of the provision of CI provision on smoking. The secondary aims are to assess the effects of ENDS and CI provision on exhaled carbon monoxide (CO), cigarette dependence, intention to quit smoking, and quitting self-efficacy, and to determine whether any changes in weight occurred secondary to the use of ENDS. Evidence of the efficacy of switching to ENDS and the use of CI could be utilized in healthcare settings to reduce the risk of morbidity and mortality among smokers with obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25 kg/m2
* smoked ≥ 5 cigarettes/day during the past year
* 21 or older
* exhaled CO of > 6 ppm at Baseline
* willing to use ENDs for 6 weeks
* daily access to a Bluetooth-enabled smartphone/tablet

Exclusion Criteria:

* planning to set a smoking quit date in the next 30 days
* receiving smoking cessation treatment of any kind in the past 30 days
* currently using ENDS > 4 day per month
* hospitalized for mental illness in past 30 days
* heart-related event (e.g., heart attack, severe angina) in past 30 days
* resides with another person enrolled in the study
* pregnant, nursing, or planning to become pregnant in the next 6 months.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Use of Cigarettes and ENDS | Assessed 4, 6, and 12 weeks follow-up
  Daily use of cigarettes and ENDS will be determined using the Timeline Follow-Back (TLFB) in follow-up assessments post-treatment.
Within-Treatment Smoking Abstinence | Daily for 4 weeks
  Number of days during the incentive period with CO verified abstinence from smoking

SECONDARY OUTCOMES:
Motivation to change | Assessed 4, 6, and 12 weeks follow-up
  Self-reported motivation, confidence, and importance of changing smoking and other tobacco & nicotine use behavior will be measured using motivation to change rulers
Carbon monoxide (CO) | Assessed 4, 6, and 12 weeks follow-up
  Exhaled breath sample used to measure carbon monoxide
Cigarette and E-Cigarette Dependence | Assessed 4, 6, and 12 weeks follow-up
  Self-reported level of dependence on cigarettes and e-cigarettes will be assessed using the Population Assessment of Tobacco and Health (PATH) Study dependence questionnaire. Items on this scale are scored from 1, "Not true of me at all", to 5, "Extremely true of me". Higher scores represent higher levels of cigarette and e-cigarette dependence. Minutes to first cigarettes daily will also be used to assess cigarette dependence with lower scores indicating greater cigarette dependence.
Comparing E-Cigarettes and Cigarettes Questionnaire | Assessed 4, 6, and 12 weeks follow-up
  Attitudes towards e-cigarettes relative to cigarettes (i.e., general benefits, general effects, and health benefits), will be assessed using the Comparing E-Cigarette and Cigarettes (CEAC) Questionnaire. Items on this questionnaire are scored from 1, "Strongly Disagree", to 5, "Strongly Agree" with higher score indicating greater agreement with benefits of e-cigarettes relative to cigarettes.
Weight | Assessed 4, 6, and 12 weeks follow-up
  Measured body weight in pounds

CONTACTS AND LOCATIONS:
Overall Officials: Cara M Murphy, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be kept and used for future research on chronic disease and substance use.
Time Frame: Clinical Laboratory Core data collected to fulfill the aims of the Center for Addiction and Disease Risk Exacerbation will be available to request immediately following publication with no prespecified end date.
Access Criteria: After all data are collected and the results of the study are published, deidentified data and biospecimens may be made available to other qualified investigators at Brown or other institutions upon request. The request will be evaluated by the investigators to ensure that it meets reasonable demands of scientific integrity.